CLINICAL TRIAL: NCT00240773
Title: A Randomized, Double-Blind, Long-Term Comparative Study Evaluating the Safety and Efficacy of Acetaminophen (4000 mg/Day) and Naproxen (750 mg/Day) in the Treatment of Osteoarthritis of the Hip or Knee
Brief Title: A Safety and Effectiveness Study of Acetaminophen (4000 mg/Day) and Naproxen (750 mg/Day) in the Treatment of Osteoarthritis of the Hip or Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002197
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: osteoarthritis hip; osteoarthritis knee; acetaminophen, naproxen
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee | interventions — Acetaminophen; Naproxen

ARMS (4):
- 001 (Experimental): acetaminophen 4 grams daily for 12 months
  Interventions: Drug: acetaminophen
- 002 (Active Comparator): naproxen 750 mg daily for 12 months
  Interventions: Drug: naproxen
- 003 (Experimental): acetaminophen 4 grams daily for six months
  Interventions: Drug: acetaminophen
- 004 (Active Comparator): naproxen 750 mg daily for six months
  Interventions: Drug: naproxen

INTERVENTIONS:
Drug: acetaminophen — 4 grams daily for six months
  Arms: 003
Drug: naproxen — 750 mg daily for 12 months
  Arms: 002
Drug: acetaminophen — 4 grams daily for 12 months
  Arms: 001
Drug: naproxen — 750 mg daily for six months
  Arms: 004

SUMMARY:
The purpose of this study is to compare the long-term safety and effectiveness of acetaminophen (4000 mg per day) and naproxen (750 mg per day) in the treatment of osteoarthritis of the hip or knee.

DETAILED DESCRIPTION:
This is a randomized, double-blind study to compare the long term safety profile and effectiveness of acetaminophen, given at a dose of 1000 mg every four to six hours, and naproxen, given at a dose of 375 mg twice daily (with matching placebo given four times daily to maintain the blind), in the treatment of osteoarthritis of the hip or knee. There are two groups of subjects. Group 1 has approximately 480 subjects randomized and a treatment duration of 12 months. Group 2 has approximately 80 subjects randomized and a treatment duration of 6 months. The primary measure of efficacy is the change from baseline in the WOMAC Osteoarthritis Index pain subscale at month 6. Safety evaluations, throughout the course of the study, include monitoring adverse events, laboratory tests and assessments of vital signs including respiration rate, pulse, blood pressure, and body weight. Subjects are instructed to take a dose of medication orally, every 4-6 hours. The acetaminophen subjects take a total daily dose of 4 g of acetaminophen. The naproxen subjects a total daily dose of 750 mg of naproxen. The treatment duration is 12 and 6 months in Group 1 and Group 2, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the hip or knee for a minimum of six months duration requiring treatment with either an analgesic or anti-inflammatory agent on a regular basis (greater than or equal to three days/week) for at least three months
* History of osteoarthritis of the hip or knee characterized by pain of mild or moderate intensity
* Radiographic evidence of grade 2 or 3 osteoarthritis based on the Kellgren and Lawrence radiographic entry criteria
* Physical ability must be either American College of Rheumatology (ACR) Functional Class I or II
* Following the washout period, reports mild to moderately severe pain over the previous 24 hours and demonstrates a minimum increase of 20% in the WOMAC Osteoarthritis Index pain subscale score, relative to the screening score.

Exclusion Criteria:

* History of surgery, including arthroscopy, or major trauma to the study joint in the previous 12 months
* Radiographic evidence of severe osteoarthritis of the study joint based on the Kellgren and Lawrence radiographic criteria of grade 4 osteoarthritis
* Signs of active study joint inflammation including redness, warmth, and/or, if qualifying with osteoarthritis of the knee, a large, bulging effusion of the study knee joint with the loss of normal contour of the joint at the screening visit or at the baseline examination after the washout period
* Morning stiffness of >30 minutes duration
* Significantly incapacitated or disabled and would be categorized as ACR Functional Class III (able to perform only few or none of the duties of usual occupation or self-care) or IV (largely or wholly incapacitated), or unable to walk without assistive devices

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the WOMAC Osteoarthritis Index pain subscale score at Month 6 or at the final visit at the time of subject discontinuation from baseline during the first six months after baseline.

SECONDARY OUTCOMES:
Change from baseline to Month 6 (or Month 12 for subjects participating in Group 1) or final visit in the WOMAC Osteoarthritis Index stiffness and physical function subscale scores.

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- See also: A Safety and Effectiveness Study of Acetaminophen (4000 mg/day) and Naproxen (750 mg/day) in the Treatment of Osteoarthritis of the Hip or Knee — http://download.veritasmedicine.com/PDF/CR002197_CSR.pdf